CLINICAL TRIAL: NCT01272024
Title: An Intervention to Improve Outcomes in Patients With Advanced Cancer
Acronym: TEAMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0909005722; R01NR011872 (NIH)
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Cancer
Keywords: clinical trial; symptom education; advanced cancer
MeSH Terms: conditions — Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Information/Education Group (Active Comparator): Assistance in using Symptom Management Toolkit
  Interventions: Behavioral: Symptom Education
- Nurse Intervention (Experimental): Participants are given intensive nurse contacts to reduce uncertainty and maximize problem solving, and later, to transition to the treatment phase of their cancer.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Symptom Education — Participants are given a Symptom Education Toolkit at baseline and at each visit thereafter (1 month and 3 month) are encouraged to use the Toolkit for symptoms they are experiencing. They are also encouraged to use resources available to them.
  Arms: Information/Education Group
Behavioral: Intervention — Participants are visited/contacted by an intervention nurse ten times over a 12-week period for the purpose of helping them to manage uncertainty and distress,to boost their problem-solving skills, and to transition to treatment.
  Arms: Nurse Intervention

SUMMARY:
1.) To integrate discharge planning into an intervention provided by advanced practice nurses (APRNs)for patients with advanced cancer, 2.) To evaluate the effects of the intervention, and 3.) To explore the reach, adoption, and implementation of the intervention to facilitate the transition of patients from surgery/biopsy/chemotherapy to medical oncology in a comprehensive cancer center.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of advanced lung, GI, Head & Neck, and Lung cancers
* post-surgical/or post-biopsy with physician's order for cancer treatment
* age 21 years or older
* lives within 50 of Yale New Haven Hospital
* has 2 or more co-morbid conditions
* has an emotional distress thermometer score of greater than or equal to 4-

Exclusion Criteria:

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2009-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Uncertainty | 1 month post baseline
  The MUIS-C contains 23 Likert scale items with scores that range from 1= strongly disagree to 5= strongly agree.
Uncertainty | 3 months post-baseline
  The MUIS-C is a 23-item scale that asks the respondent to rate items on a scale of 1=strongly disagree to 5= strongly agree.

SECONDARY OUTCOMES:
HADS- Anxiety | 1 month post baseline
  7 items are rated on a 4-point scale.
HADS-Anxiety | 3 months post baseline.
  7 items are rated on a 4-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth McCorkle, RN, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital/Smilow Cancer Hospital, New Haven, Connecticut, United States